CLINICAL TRIAL: NCT07331688
Title: CMTS0515 - Augmented Washed Microbiota Transplantation Versus Washed Microbiota Transplantation in Radiation Enteritis: A Randomized, Double-Blind, Non-inferiority Trial
Brief Title: CMTS0515-auWMT for Radiation Enteritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WMT-CMTS0515-RE
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Radiation Enteritis
Keywords: Fecal Microbiota Transplantation; Washed Microbiota Transplantation; Radiotherapy; Radiation Enteritis; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMTS0515-augmented washed microbiota transplantation (Experimental): Patients undergo CMTS0515-augmented washed microbiota transplantation once a day for three consecutive days.
  Interventions: Other: CMTS0515-augmented washed microbiota transplantation
- washed microbiota transplantation (Active Comparator): Patients undergo washed microbiota transplantation once a day for three consecutive days.
  Interventions: Other: Washed Microbiota Transplantation

INTERVENTIONS:
Other: CMTS0515-augmented washed microbiota transplantation — Lyophilized CMTS0515 is added to washed microbiota suspension and administered via mid-gut or colonic transendoscopic enteral tube.
  Arms: CMTS0515-augmented washed microbiota transplantation
Other: Washed Microbiota Transplantation — Washed microbiota suspension delivered through mid-gut and lower-gut transendoscopic enteral tube.
  Arms: washed microbiota transplantation

SUMMARY:
This is a randomized controlled trial to explore the exploring the non-inferiority of CMTS0515-augmented WMT compared to WMT.

DETAILED DESCRIPTION:
At least 60 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. They will be randomly assigned to the experimental group (CMTS0515-augmented WMT) and the control group (WMT). Data of demographic characteristics, intestinal symptoms, medicine treatment usage and clinical outcomes will be collected. After treatment, they will enter the follow-up period for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of abdominal or pelvic cancer;
2. Completion of at least one entire course of radiation therapy;
3. Age ≥18 years at the time of cancer diagnosis.

Exclusion Criteria:

1. Absence of intestinal symptoms or transient intestinal symptoms;
2. Radiation treatment involving areas outside the abdomen and pelvis;
3. Diagnosis of antibiotic-associated diarrhea or use of antibiotics within four weeks before enrollment;
4. Presence of intestinal comorbidities, including inflammatory bowel disease or pseudomembranous colitis;
5. Presence of severe conditions rendering the patient unsuitable for inclusion;
6. Experience of bowel surgery for RE-associated fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The clinical response rate after treatment | 1 week, 4 weeks and 8 weeks
  Radiation Therapy Oncology Group (RTOG) scores

SECONDARY OUTCOMES:
Scores of gastrointestinal symptoms | 1 week, 4 weeks and 8 weeks
  Gastrointestinal symptoms will be evaluated according to NCI-CTC 5.0
Stool frequency and consistency | 1 week, 4 weeks and 8 weeks
  Stool frequency and consistency will be evaluated according to The Bristol Stool Form Scale (BSFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Microbiota Medicine & Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China